CLINICAL TRIAL: NCT02219243
Title: Modification of Interpretive Biases in Children With Social Anxiety
Brief Title: Interpretive Biases in Children With Social Anxiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Han Joo Lee, Assistant Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWM14.141
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Social Anxiety; Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Cognitive Training; Interpretation Modification Program
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Waitlist Control (No Intervention): This is a 1-month waitlist control to be compared with the active online interpretation training interventions. This is a no intervention control group
- Active Interpretation Training (Experimental): Online Interpretation Training Condition 2 provides three sessions of a computerized training. Each session will last approximately 20-30 minutes, and participants will undergo 1 session each week.
  Interventions: Behavioral: Online Interpretation Training Condition 1
- Placebo Interpretation Training (Experimental): Online Interpretation Training Condition 1 provides three sessions of a computerized training. Each session will last approximately 20-30 minutes, and participants will undergo 1 session each week.
  Interventions: Behavioral: Online Interpretation Training Condition 2

INTERVENTIONS:
Behavioral: Online Interpretation Training Condition 1 — The online computerized training is a web-based tool that modifies how children interpret ambiguous scenarios.
  Arms: Active Interpretation Training
Behavioral: Online Interpretation Training Condition 2 — The online computerized training is a web-based tool that modifies how children interpret ambiguous scenarios.
  Arms: Placebo Interpretation Training

SUMMARY:
A substantial number of children with social anxiety fail to gain benefit from contemporary cognitive-behavior therapy (CBT) approaches. More novel treatment approaches for treatment of social anxiety are needed. The current study attempts to modify an interpretation style that is characteristic of children who also display high anxiety in social situations. Participants between the ages of 8-12 years old, with social anxiety, will be randomly assigned to one of three treatment conditions: two conditions are designed to manipulate the interpretation bias or a wait-list control condition. All study procedures will be conducted online. This study will help develop an effective cognitive intervention program for social anxiety in children.

DETAILED DESCRIPTION:
The current study aims to test the effectiveness of computer-based interpretation bias modification training as a therapeutic intervention for social anxiety disorder (SAD). Individuals who experience social anxiety often have difficulty in engaging in social situations, such as speaking in front of a group and maintaining a conversation. For youngsters, this may take the form of avoidance, including avoiding situations such as raising one's hand in class, eating in front of other people and participating in small group activities. Additionally, those with social anxiety are more likely to interpret ambiguous social scenarios in a threatening way than are control subjects (Bogels, Snieder, & Kindt, 2003; Miers, Blote, Bogels, & Westenberg, 2008; Vassilopoulos & Banerjee, 2008; Vassilopoulos, 2006; Muris, Meckelbach, & Damsma, 2000). Research has shown that interpretation biases are modifiable at a young age (Muris, Huijding, Mayer, & Hameetman, 2008; Vassilopoulous, Bangerjee, Prantzalou, 2009; Muris, Huijding, Mayer, Remmerswaal, & Vreden, 2009; Lothmann, Holmes, Chan, & Lau, 2010).

Participants between the ages of 8-12 years old, with social anxiety, will be randomly assigned to one of three treatment conditions: two conditions are designed to manipulate the interpretation bias or a wait-list control condition. All study procedures will be conducted online. Subjects do not need to come to the University of Wisconsin-Milwaukee to participate. Thirty children with social anxiety will be randomly assigned to one of the three conditions, and will be assessed at baseline, post-treatment, and 1-month follow-up. The waitlisted participants will also be invited to undergo the training program after the 1-month follow-up assessment is completed. This study is expected to generate important data that will guide the development of an accessible, cost-efficient, and effective cognitive intervention for individuals suffering from social anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 8-12
* Diagnosis of social anxiety disorder
* Overall IQ score of 80 or greater
* Speak English fluently as the primary language
* Working internet connection with access to Skype or Facetime video conferencing software

Exclusion Criteria:

* Attention Deficit Hyperactivity Disorder, Oppositional Defiant Disorder or Conduct Disorder
* Pervasive developmental disorder or autism-spectrum disorder
* Past or active psychosis, bipolar disorder, or schizophrenia
* Current evidence-based cognitive-behavioral treatment for social anxiety problems
* Past cognitive behavioral treatment for social anxiety problems that lasted at least 3 sessions
* Significant suicidal ideation and/or attempts within the past 3 months
* Any recent (within the past 4 weeks) or planned changes in medication
* Reading disorder or impairments in reading ability.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change on the Liebowitz Social Anxiety Scale for Children and Adolescents | Baseline, 4-weeks, and 1-month follow-up
  A clinician-rated measure for assessing the severity of social anxiety and the impairment caused by it. This measure will be administered at baseline, at 4 weeks, and at 1-month follow-up.

SECONDARY OUTCOMES:
Change on the Multidimensional Anxiety Scale for Children-2nd edition Parent and Self Report | Baseline, 4 weeks, and 1-month Follow-up
  This is a widely used assessment tool for symptoms of anxiety disorders. This measure will be administered at baseline, at 4 weeks, and at 1-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- UWM Anxiety Disorders Laboratory, Milwaukee, Wisconsin, United States